CLINICAL TRIAL: NCT00179777
Title: TRIGR - Trial to Reduce IDDM in the Genetically at Risk
Brief Title: TRIGR - Primary Prevention Study for Type 1 Diabetes in Children at Risk
Acronym: TRIGR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: United States Congress (U.S. Federal Agency); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); Juvenile Diabetes Research Foundation (Other); European Community (EC) (Other Government); European Foundation for the Study of Diabetes (Other); Mead Johnson Nutrition (Industry); Academy of Finland (Other); Diabetes Research Foundation, Finland (Other); Dutch Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Mikael Knip, Professor, Principal Investigator, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MCT-49395; U01HD040364 (NIH); U01HD042444 (NIH)
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Results first posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Genetic Predisposition to Disease; Infant Nutrition; Primary Prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Genetic Predisposition to Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrolysed infant formula (Experimental): Hydrolysed infant formula
  Interventions: Dietary Supplement: Hydrolysed infant formula
- Nonhydrolysed infant formula (Placebo Comparator): Nonhydrolysed cow's milk based infant formula
  Interventions: Dietary Supplement: Nonhydrolysed infant formula

INTERVENTIONS:
Dietary Supplement: Hydrolysed infant formula — Participants in the Hydrolysed infant formula -group received the test formula, casein hydrolysate (Nutramigen™, Mead Johnson Nutritionals), not containing antigenic CM protein, whenever breast milk is not available.
  Arms: Hydrolysed infant formula
Dietary Supplement: Nonhydrolysed infant formula — Participants in the Nonydrolysed infant formula -group received the CM protein containing control formula which has an addition (20 %) of Nutramigen, whenever breast milk is not available.
  Arms: Nonhydrolysed infant formula

SUMMARY:
The Trial to Reduce IDDM in the Genetically at Risk (TRIGR) is an international effort to conduct a primary prevention nutrition trial for type 1 (insulin-dependent) diabetes. The TRIGR study was targeted at newborns who are at genetic risk for type 1 diabetes because their mother, father and/or full sibling has type 1 diabetes. All families were encouraged to breast feed their infants for as long as possible. Prior to birth, the child was randomly assigned to receive one of two infant formulas, should formula be required prior to 8 months of age. The study determined whether weaning to a possibly protective infant formula decreases these children's chances of developing diabetes - as it does in the animal models for diabetes.

DETAILED DESCRIPTION:
The hypothesis for this study is that weaning to an extensively hydrolyzed infant formula will decrease the incidence of type 1 diabetes in subjects with risk-associated HLA genotypes and a first degree relative with type 1 diabetes, as it does in all relevant animal models for the disease.

Specific Aims:

I.a: To determine if weaning to a casein hydrolysate infant formula reduces the frequency of diabetes-predictive auto-antibodies in subjects with risk-associated HLA genotype and a first degree relative with type 1 diabetes (mother, father and/or full sibling).

I-b: To determine if weaning to a casein hydrolysate infant formula reduces the frequency of clinical diabetes in subjects with risk-associated HLA genotype and an affected first degree relative.

A secondary aim is to determine relationships between cow's milk antibodies, a measure of cow's milk exposure, and diabetes-associated auto-antibodies.

The mother of the unborn child is recruited during pregnancy. Randomization to one of two infant formulas takes place before birth (after 35 weeks gestation) or immediately after birth.

Experimental Arm: Use of extensively hydrolysed cow's milk based infant formula when needed in supplementation or substitution for breast milk through 6-8 months from birth.

Control Arm: Use of non-hydrolysed cow's milk based infant formula when needed in supplementation or substitution for breast milk through 6-8 months from birth.

All families were encouraged to breast feed their infants for as long as possible. The study infant formula was only used if exclusive breast feeding ceases before 8 months of age.

Cord blood for genotyping was obtained at birth, or failing that from a heel prick by 7 days of age. Only subjects with genotypes indicating increased genetic risk for type 1 diabetes remained in the intervention trial. All other subjects were withdrawn from the study.

All subjects were followed until the youngest subject turns age 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Biological parent and/or full (not half) sibling of the newborn infant had type 1 diabetes as defined by the World Health Organization
* The infant's parent or legal guardians gave signed consent to participate

Exclusion Criteria:

* An older sibling of the newborn infant had been included in the TRIGR intervention
* Multiple gestation
* The parents were unwilling or unable to feed the infant cow's milk based products for any reason (e.g., religious, cultural).
* The newborn infant had a recognizable severe illness such as those due to chromosomal abnormality, congenital malformation, respiratory failure needing assisted ventilation, enzyme deficiencies, etc.
* The gestational age of the newborn infant was less than 35 weeks.
* The infant was older than 7 days at randomization.
* Inability of the family to take part in the study (e.g. the family has no access to any of the Study Centers, the family has no telephone).
* The infant had received any infant formula other than Nutramigen prior to randomization.
* No HLA sample drawn before the age of 8 days.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5156 (Actual)
Dates: Start 2002-05-06 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Knip, MD, Principal Investigator — University of Helsinki
Locations (18):
- United States (2):
  - The University of South Florida, Tampa, Florida
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Children's Hospital at Westmead, Westmead, New South Wales, Australia
- Robarts Research Institute, London, Ontario, Canada
- 3rd Faculty of Medicine, Charles University, University Hospital Vinohrady, Prague, Czechia
- Tartu University Children's Hospital, Tartu, Estonia
- University of Helsinki, Helsinki, Finland
- Kinderkrankenhaus auf der Bult, Hanover, Germany
- Semmelweis Medical University, Budapest, Hungary
- Italy (2):
  - St. Michele Hospital, Cagliari, Sardinia
  - University Campus Bio-Medico of Rome, Rome
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Sophia Children's Hospital, Rotterdam, Netherlands
- Medical University of Wroclaw, Wroclaw, Poland
- Spain (2):
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital Clinico San Carlos, Madrid
- University of Linkoping, Linköping, Sweden
- University Children's Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akerblom HK, Virtanen SM, Ilonen J, Savilahti E, Vaarala O, Reunanen A, Teramo K, Hamalainen AM, Paronen J, Riikjarv MA, Ormisson A, Ludvigsson J, Dosch HM, Hakulinen T, Knip M; National TRIGR Study Groups. Dietary manipulation of beta cell autoimmunity in infants at increased risk of type 1 diabetes: a pilot study. Diabetologia. 2005 May;48(5):829-37. doi: 10.1007/s00125-005-1733-3. Epub 2005 Apr 19. PMID 15838685
- [Background] TRIGR Study Group. Study design of the Trial to Reduce IDDM in the Genetically at Risk (TRIGR). Pediatr Diabetes. 2007 Jun;8(3):117-37. doi: 10.1111/j.1399-5448.2007.00239.x. PMID 17550422
- [Background] Åkerblom HK, Knip M, Becker D, Dosch H-M, Dupré J, Ilonen J, Krischer JP and the TRIGR Study Group. The TRIGR Trial: Testing the Potential Link between Weaning Diet and Type 1 Diabetes. Immun, Endoc, Metab Agents in Med Chem 7:251-263, 2007.
- [Result] Writing Group for the TRIGR Study Group; Knip M, Akerblom HK, Al Taji E, Becker D, Bruining J, Castano L, Danne T, de Beaufort C, Dosch HM, Dupre J, Fraser WD, Howard N, Ilonen J, Konrad D, Kordonouri O, Krischer JP, Lawson ML, Ludvigsson J, Madacsy L, Mahon JL, Ormisson A, Palmer JP, Pozzilli P, Savilahti E, Serrano-Rios M, Songini M, Taback S, Vaarala O, White NH, Virtanen SM, Wasikowa R. Effect of Hydrolyzed Infant Formula vs Conventional Formula on Risk of Type 1 Diabetes: The TRIGR Randomized Clinical Trial. JAMA. 2018 Jan 2;319(1):38-48. doi: 10.1001/jama.2017.19826. PMID 29297078
- [Derived] Biradar R, Kalim UU, Lonnberg T, Junttila S, Suomi T, Norman SZ, Starskaia I, Paulin N, Mikkola L, Vaarala O, Rasool O, Knip M, Elo LL, Lahesmaa R. Single-cell RNA-seq analysis of longitudinal CD4+ T cell samples reveals cell-type-specific changes during early stages of type 1 diabetes. Genome Med. 2025 Dec 29;17(1):154. doi: 10.1186/s13073-025-01574-x. PMID 41462339
- [Derived] Niinisto S, Cuthbertson D, Miettinen ME, Hakola L, Nucci A, Korhonen TE, Hyoty H, Krischer JP, Vaarala O, Knip M, Savilahti E, Virtanen SM; TRIGR Investigators. High Concentrations of Immunoglobulin G Against Cow Milk Proteins and Frequency of Cow Milk Consumption Are Associated With the Development of Islet Autoimmunity and Type 1 Diabetes-The Trial to Reduce Insulin-dependent Diabetes Mellitus (IDDM) in the Genetically at Risk (TRIGR) Study. J Nutr. 2024 Aug;154(8):2493-2500. doi: 10.1016/j.tjnut.2024.06.005. Epub 2024 Jun 19. PMID 38906178
- [Derived] Niinisto S, Miettinen ME, Cuthbertson D, Honkanen J, Hakola L, Autio R, Erlund I, Arohonka P, Vuorela A, Harkonen T, Hyoty H, Krischer JP, Vaarala O, Knip M, Virtanen SM; TRIGR Investigators. Associations Between Serum Fatty Acids and Immunological Markers in Children Developing Islet Autoimmunity-The TRIGR Nested Case-Control Study. Front Immunol. 2022 May 25;13:858875. doi: 10.3389/fimmu.2022.858875. eCollection 2022. PMID 35693790
- [Derived] Nucci AM, Virtanen SM, Cuthbertson D, Ludvigsson J, Einberg U, Huot C, Castano L, Aschemeier B, Becker DJ, Knip M, Krischer JP; TRIGR Investigators. Growth and development of islet autoimmunity and type 1 diabetes in children genetically at risk. Diabetologia. 2021 Apr;64(4):826-835. doi: 10.1007/s00125-020-05358-3. Epub 2021 Jan 21. PMID 33474583
- [Derived] Pacaud D, Nucci AM, Cuthbertson D, Becker DJ, Virtanen SM, Ludvigsson J, Ilonen J, Knip M; TRIGR investigators. Association between family history, early growth and the risk of beta cell autoimmunity in children at risk for type 1 diabetes. Diabetologia. 2021 Jan;64(1):119-128. doi: 10.1007/s00125-020-05287-1. Epub 2020 Oct 7. PMID 33026463
- [Derived] Krischer JP, Cuthbertson D, Couluris M, Knip M, Virtanen SM. Association of diabetes-related autoantibodies with the incidence of asthma, eczema and allergic rhinitis in the TRIGR randomised clinical trial. Diabetologia. 2020 Sep;63(9):1796-1807. doi: 10.1007/s00125-020-05188-3. Epub 2020 Jun 17. PMID 32548702
- [Derived] Miettinen ME, Niinisto S, Erlund I, Cuthbertson D, Nucci AM, Honkanen J, Vaarala O, Hyoty H, Krischer JP, Knip M, Virtanen SM; TRIGR Investigators. Serum 25-hydroxyvitamin D concentration in childhood and risk of islet autoimmunity and type 1 diabetes: the TRIGR nested case-control ancillary study. Diabetologia. 2020 Apr;63(4):780-787. doi: 10.1007/s00125-019-05077-4. Epub 2020 Jan 7. PMID 31912198
- [Derived] Knip M, Akerblom HK, Becker D, Dosch HM, Dupre J, Fraser W, Howard N, Ilonen J, Krischer JP, Kordonouri O, Lawson ML, Palmer JP, Savilahti E, Vaarala O, Virtanen SM; TRIGR Study Group. Hydrolyzed infant formula and early beta-cell autoimmunity: a randomized clinical trial. JAMA. 2014 Jun 11;311(22):2279-87. doi: 10.1001/jama.2014.5610. PMID 24915259
- [Derived] Franciscus M, Nucci A, Bradley B, Suomalainen H, Greenberg E, Laforte D, Kleemola P, Hyytinen M, Salonen M, Martin MJ, Catte D, Catteau J; TRIGR Investigators. Recruitment and retention of participants for an international type 1 diabetes prevention trial: a coordinators' perspective. Clin Trials. 2014 Apr;11(2):150-8. doi: 10.1177/1740774513510070. Epub 2013 Nov 11. PMID 24216218
- [Derived] TRIGR Study Group; Akerblom HK, Krischer J, Virtanen SM, Berseth C, Becker D, Dupre J, Ilonen J, Trucco M, Savilahti E, Koski K, Pajakkala E, Fransiscus M, Lough G, Bradley B, Koski M, Knip M. The Trial to Reduce IDDM in the Genetically at Risk (TRIGR) study: recruitment, intervention and follow-up. Diabetologia. 2011 Mar;54(3):627-33. doi: 10.1007/s00125-010-1964-9. Epub 2010 Dec 12. PMID 21153533
- See also: TRIGR International website - Click here for more information on this study - www.TRIGR.org — https://www.trigr.org
- See also: TRIGR North America website - Click here for more information on this study - www.trigrnorthamerica.org — http://www.trigrnorthamerica.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2002-2007 Recruited through local clinics and obstetrics unit
Groups:
- Hydrolysed Infant Formula: Hydrolysed infant formula
  hydrolysed infant formula: hydrolysed infant formula
- Nonhydrolysed Infant Formula: Nonhydrolysed infant formula
  nonhydrolysed infant formula: nonhydrolysed infant formula
Period: Overall Study
Arm/Group | Hydrolysed Infant Formula | Nonhydrolysed Infant Formula
Started | 2613 | 2543
Completed | 1081 | 1078
Not Completed | 1532 | 1465

BASELINE CHARACTERISTICS:
Population: Analysis population consisted of participants with increased genetic risk (defined HLA genotypes) for type 1 diabetes.
Groups:
- Nonhydrolysed Infant Formula: A conventional adapted cow's milk formula supplemented with 20% of the casein hydrolysate.
- Hydrolysed Infant Formula: Hydrolysed Infant Formula missing intact cows milk proteins
- Total: Total of all reporting groups
Arm/Group | Nonhydrolysed Infant Formula | Hydrolysed Infant Formula | Total
Number analyzed (Participants) | 1078 | 1081 | 2159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1078 | 1081 | 2159
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] — Age at Randomization and Last Follow-up, years
  years
    At at randomization | 0 [0 to 0] | 0 [0 to 0] | 0 [0.0 to 0.0]
    Age at Last Follow-up | 11.96 [0.07 to 15.61] | 11.93 [0.24 to 15.29] | 11.95 [0.07 to 15.61]
Sex: Female, Male [Count of Participants; unit: Participants] — Sex (female, male) of the participants
  Participants
    Female | 516 | 505 | 1021
    Male | 562 | 576 | 1138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethicity, reported on the Study Registration form, information received from the parents
  Participants
    Hispanic or Latino | 53 | 53 | 106
    Not Hispanic or Latino | 987 | 989 | 1976
    Unknown or Not Reported | 38 | 39 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race reported on the Study Registration form, information received form the parents
  Participants
    American Indian or Alaska Native | 3 | 3 | 6
    Asian | 10 | 13 | 23
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 10 | 16 | 26
    White | 1040 | 1034 | 2074
    More than one race | 9 | 6 | 15
    Unknown or Not Reported | 6 | 9 | 15
Region of Enrollment [Number; unit: participants] — Region of Enrollments by Country, information based on registration
  participants
    Hungary | 12 | 11 | 23
    United States | 196 | 199 | 395
    Czechia | 82 | 82 | 164
    Switzerland | 6 | 37 | 43
    Spain | 31 | 29 | 60
    Canada | 262 | 265 | 527
    Netherlands | 29 | 24 | 53
    Sweden | 47 | 49 | 96
    Luxembourg | 3 | 4 | 7
    Finland | 212 | 212 | 424
    Poland | 46 | 48 | 94
    Italy | 26 | 28 | 54
    Australia | 51 | 51 | 102
    Germany | 57 | 55 | 112
    Estonia | 18 | 17 | 35
family history of type 1 diabetes [Count of Participants; unit: Participants] — Family History of Type 1 Diabetes (mother, father or sibling had Type 1 diabetes), information received from the parents
  Participants
    Only mother with type 1 diabetes | 522 | 530 | 1052
    Only father with type 1 diabetes | 367 | 355 | 722
    Only one sibling with type 1 diabetes | 157 | 151 | 308
    More than one family member with type 1 diabetes | 32 | 45 | 77

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Type 1 Diabetes Mellitus
Description: Number of participants with Type 1 diabetes mellitus assessed by (1) blood glucose and HbA1c at 12 and 18 months of age, and annually from age 2 to 10 years, and (2) oral glucose tolerance test at 6 and 10 years of age and in the final year of the study.
Time Frame: 12 and 18 months and annually from 2 years up to 14 years
Population: Analysis population consisted of participants with increased genetic risk (defined HLA genotypes) for type 1 diabetes
Measure: Number; unit: participants
Groups:
- Nonhydrolysed Infant Formula; Hydrolysed Infant Formula: Number of participants diagnosed with type 1 diabetes
Arm/Group | Nonhydrolysed Infant Formula | Hydrolysed Infant Formula
Number analyzed (Participants) | 1078 | 1081
participants | 82 | 91

2. Secondary Outcome: Number of Participants With Diabetes Associated Autoantibodies
Description: Diabetes associated autoantibodies (ICA, IAA, GADA, IA-2A) at 3, 6, 9, 12, and 18 months of age, and annually from age 2 to 10-14 years
Time Frame: 3, 6, 9, 12, 18 months and annually from 2 years up to 14 years
Population: Analysis population consisted of participants with increased genetic risk (defined HLA genotypes) for type 1 diabetes
Measure: Count of Participants; unit: Participants
Groups:
- Nonhydrolysed Infant Formula: Diabetes associated autoantibodies (ICA, IAA, GADA, IA-2A) in the nonhydrolysed infant formula
- Hydrolysed Infant Formula: Diabetes associated autoantibodies (ICA, IAA, GADA, IA-2A) in the hydrolysed infant formula
Arm/Group | Nonhydrolysed Infant Formula | Hydrolysed Infant Formula
Number analyzed (Participants) | 1078 | 1081
Participants
  ICA+ | 373 | 394
  IAA+ | 162 | 183
  GADA+ | 186 | 207
  IA-2A+ | 102 | 115

ADVERSE EVENTS:
Time Frame: 11.5 years
Groups:
- Nonhydrolysed Infant Formula: Reported Adverse Events during the Follow-up in the Nonhydrolysed Infant Formula Group
- Hydrolysed Infant Formula: Reported Adverse Events during the Follow-up in the Hydrolysed Infant Formula Group
Arm/Group | Nonhydrolysed Infant Formula | Hydrolysed Infant Formula
All-Cause Mortality (participants affected / at risk) | 5/1078 | 5/1081
Serious Adverse Events (participants affected / at risk) | 379/1078 | 377/1081
Other Adverse Events (participants affected / at risk) | 1010/1078 | 1012/1081
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nonhydrolysed Infant Formula (N=1078) | Hydrolysed Infant Formula (N=1081)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 51 (64) | 46 (56)
Gastroenteritis (Gastrointestinal disorders) | 35 (46) | 29 (36)
Urinary Tract Infection (Renal and urinary disorders) | 12 (12) | 11 (13)
Middle Ear Infection (Ear and labyrinth disorders) | 23 (24) | 27 (35)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 9 (9)
Other Unspecified Infection (Infections and infestations) | 62 (64) | 61 (65)
Suspected Study Formula Intolerence (Gastrointestinal disorders) | 5 (5) | 3 (3)
Asthma, Other Forms of Allergy (Respiratory, thoracic and mediastinal disorders) | 10 (14) | 15 (15)
Malignancy (General disorders) | 1 (1) | 2 (2)
Accident (Not Requiring Hospitalization) (General disorders) | 9 (11) | 11 (13)
Accident (Requiring Hospitalization) (General disorders) | 27 (29) | 23 (25)
Hospitalization (General disorders) | 47 (58) | 52 (75) — Event requiring inpatient hospitalization or prolongation of existing hospitalization
Life-threatening event (General disorders) | 4 (4) | 2 (2)
Disability/incapacity (Injury, poisoning and procedural complications) | 3 (3) | 1 (2) — Persistent or significant disability/incapacity
Other Unspecified Adverse Event (General disorders) | 190 (268) | 215 (320)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nonhydrolysed Infant Formula (N=1078) | Hydrolysed Infant Formula (N=1081)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 772 (6206) | 754 (5952)
Gastroenteritis (Gastrointestinal disorders) | 515 (1519) | 494 (1598)
Urinary Tract Infection (Renal and urinary disorders) | 91 (123) | 80 (130)
Middle Ear Infection (Ear and labyrinth disorders) | 534 (1951) | 525 (1796)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 93 (119) | 91 (110)
Other, unspecified infection (Infections and infestations) | 765 (3285) | 740 (3226)
Suspected Study Formula Intolerance (Gastrointestinal disorders) | 56 (73) | 49 (61)
Asthma, other forms of allergy (Respiratory, thoracic and mediastinal disorders) | 359 (783) | 332 (696)
Accident, not requiring hospitalization (Injury, poisoning and procedural complications) | 151 (194) | 140 (189)
Hypoglycemia requiring IV glucose (Endocrine disorders) | 20 (20) | 10 (10)
Other, unspecified adverse event (General disorders) | 804 (4452) | 814 (4380)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT00179777/Prot_SAP_000.pdf